CLINICAL TRIAL: NCT02897206
Title: Imipenem Prophylaxis of Infectious Complications in Patients With Acute Pancreatitis
Brief Title: Imipenem Prophylaxis in Patients With Acute Pancreatitis
Acronym: IMPROWE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Rijeka (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Principal Investigator, Goran Poropat, Postdoctoral Researcher, University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13.06.1.2.30
Record Dates: First submitted 2015-12-20; First posted 2016-09-13 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis; Antibiotic prophylaxis; Imipenem-cilastatin; Infected pancreatic necrosis; Infection; Organ failure
MeSH Terms: conditions — Pancreatitis; Infections | interventions — Imipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imipenem group (Experimental): Imipenem 3 x 500 mg i.v. daily ideally for 10 days (minimum 7 days, maximum 21 days)
  Interventions: Drug: Imipenem
- Placebo group (Placebo Comparator): Identical placebo administered in identical dosage, timing and duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imipenem — A wide-spectre antibiotic from the carbapenem group
  Other Names: Imipenem-cilastatin
  Arms: Imipenem group
Drug: Placebo — An imipenem-matching placebo
  Arms: Placebo group

SUMMARY:
This is a prospective, single-center, randomized, placebo-controlled, double-blind clinical trial that aims to investigate the beneficial and harmful effects of prophylactic use of imipenem in patients with predicted severe acute pancreatitis. All patients with first attack of acute pancreatitis, an onset of disease less than 72h before admission, and an APACHE II score ≥ 8 calculated within the first 24h from admission will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute pancreatitis defined by the Revised 2012 Atlanta Criteria
* first manifestation of acute pancreatitis regardless of etiology
* APACHE II ≥ 8 calculated within the first 24 hours of admission
* onset of symptoms < 72 hours before admission

Exclusion Criteria:

* age < 18 years
* pregnant and breastfeeding women
* active and documented infection at admission
* concomitant antibiotic treatment or antibiotic treatment present within 72 hours before enrollment
* acute pancreatitis diagnosed at surgery
* active malignancy
* known immune deficiency
* patients with chronic pancreatitis
* patients unwilling to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Infectious complications | 30 days

SECONDARY OUTCOMES:
Mortality | 30 days
Number of patients with Systemic Inflammatory Response Syndrome (SIRS) | 30 days
  SIRS was defined as presence of at least two following parameters for a continuous period of ≥ 48 hours: body temperature >38°C or <36°C; heart rate >90 beats per minute; hyperventilation with a respiratory rate >20 breath per minute or a PaCO2 < 32 mmHg; and white blood cell count >12000/mm3 or <4000/mm3.
Local complications | 30 days
Systemic complications | 30 days
Number of patients with persistent and transitory organ failure (cardiovascular, respiratory, renal) | 30 days
  Marshall organ dysfunction scoring system (MODS) was used to define organ failure in the case of cardiovascular, renal and respiratory system function.
Surgical interventions | 30 days
  The investigators will register the number of patients requiring surgical interventions for acute pancreatitis.
Serious adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Davor Stimac, MD, PhD, Principal Investigator — Department of Gastroenterology, University Hospital Rijeka
Locations (1):
- University Hospital Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poropat G, Radovan A, Peric M, Mikolasevic I, Giljaca V, Hauser G, Milic S, Stimac D. Prevention of Infectious Complications in Acute Pancreatitis: Results of a Single-Center, Randomized, Controlled Trial. Pancreas. 2019 Sep;48(8):1056-1060. doi: 10.1097/MPA.0000000000001368. PMID 31404018